CLINICAL TRIAL: NCT03165552
Title: An Educational Intervention to Prevent Acute Kidney Injury in Primary Care. The ED-AKI-P Implementation Study
Acronym: ED-AKI-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0524
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Educational Arm (Experimental): This group will receive an acute kidney injury educational intervention
  Interventions: Other: Acute kidney injury education

INTERVENTIONS:
Other: Acute kidney injury education — A face to face, a constructivist learning approach to encourage users to explore and learn about the topic of AKI in a way that maximises educational value. The programme is supported by a web based resource that presents a series of realistic case studies highlighting common causes of AKI in primary care designed to be easy to access and navigate, whilst being visual and interactive to enhance user engagement. The educayion is delivered to healthcare staff not to patients.

SUMMARY:
Patients with abnormal kidney function are common in primary care, particularly in people with other long standing illnesses. Some of these patients have long standing weakness of their kidneys, others develop new kidney weakness alongside other new illnesses. Patients with weak kidneys are more likely to be admitted to hospital, spend longer in hospital or die than those with normal kidneys. Although these events are common, how kidney weakness develops in the community is not well understood and awareness is poor. It is known that appropriate attention to a patient's medical care at times of high risk may reduce the onset of new kidney weakness. We have developed a new education package for primary healthcare professionals and patients. This will teach them about risks of new kidney weakness in their patients, give advice about how to combat them, and help prevent it occurring. This project will also use a new software tool - IMPAKT EVOLVE-AKI - to extract information from primary care systems and combine this with hospital data to identify developing kidney weakness much more accurately primary care . Both these elements of the study have already been tested in primary care and we are confident that they work well. Patients and the public have been involved in the development of these tools and will also be closely involved in their implementation. We now intend to implement the education more widely in primary care. We will then test how effectively the education has been implemented and whether it has a significant effect on the number of episodes of new kidney weakness developing in primary care. We calculate that we will need to provide this education to 36 practices to be able to determine accurately whether the programme significantly reduces new kidney weakness. Advice we have received from colleagues in primary care indicates that they are very interested in this education programme, and we believe that that a positive result from this study will lead to rapid and wide implementation of this combined programme of education and data analysis to the benefit of patients across the UK. This study fits well with a national programme of work in this area, and this combination will help with wider adoption of the study findings when the results are available.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common cause of excess morbidity and mortality amongst patients with long term conditions, and is a common finding in patients admitted acutely into hospital. Although the disease commonly develops in the community there is little evidence to guide identification of patients at risk or how best to educate healthcare workers in primary care to improve the care of patients at risk of AKI. We hypothesise firstly that: an AKI educational intervention in primary care can be delivered to healthcare practitioners with high integrity, and secondly that: an AKI educational intervention delivered in primary care will result in a decreased incidence of AKI in the community. To test this we will build on pilot work that detects high-AKI risk patients and provides education for healthcare workers and at-risk patients. The study will bring together novel informatics, and education programme for primary healthcare workers along with patient information and guidance. Recruitment will be at the practice level and will take place after the delivery of the face to face educational intervention. Recruited practices will have their high risk AKI patients identified using web based software, and GPs will be encouraged, where clinically appropriate, to contact patients with an educational leaflet advising them how to prevent AKI by stopping medications under certain circumstances. In addition a variety of associated biomedical data will be obtained from practice IT systems to identify the preceding incidence of AKI in any recruited practice. Eighteen months after the delivery of the education intervention the incidence of AKI in each practice will again be determined to examine the effect of the educational intervention on AKI incidence. The fidelity of delivery of the education intervention will also be studied using qualitative techniques. Power calculations suggest that 36 practices will need to participate to detect a 25% reduction in AKI incidence. We anticipate that this programme will effectively reduce AKI community incidence and will be of significant interest to commissioners. Study findings will be disseminated through a variety of avenues including through structures established by NHS England to support improvements in AKI management.

ELIGIBILITY:
Inclusion criteria:

All patients aged over 18 registered with the practice

Exclusion criteria:

Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury before and after educational intervention | 18 months
  The incidence of AKI in a group of practices will be measured before and after an educational intervention